CLINICAL TRIAL: NCT07115992
Title: Efficacy and Safety of Radical Prostatectomy (RP) With or Without Salvage Radiotherapy Versus RP With Extended Pelvic Lymph Node Dissection for Localized Intermediate- and High-risk Prostate Cancer With a Briganti Nomogram≥7%: an Open-label, Single-center, Non-inferiority Randomized Controlled Study
Brief Title: Efficacy and Safety of Radical Prostatectomy (RP) With or Without Salvage Radiotherapy Versus RP With Extended Pelvic Lymph Node Dissection for Localized Intermediate- and High-risk Prostate Cancer With a Briganti Nomogram≥7%
Acronym: PRESEL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-423
Record Dates: First submitted 2025-07-24; First posted 2025-08-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Prostate Adenoma
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will receive robot-assisted laparoscopic radical prostatectomy (RARP), followed by salvage radiotherapy only if biochemical recurrence occurs postoperatively.
  Interventions: Procedure: RARP±SRT
- Control group (Active Comparator): Participants in the control group will receive RARP with extended pelvic lymph node dissection, per guideline recommendations.
  Interventions: Procedure: RARP+ePLND

INTERVENTIONS:
Procedure: RARP±SRT — Participants will undergo robot-assisted radical prostatectomy (RARP). Upon biochemical recurrence, they will receive salvage radiotherapy: 52.5-62.5 Gy in 20-25 fractions/2.5-3.0 Gy per fraction, per 2025 AUA/ASTRO/SUO guidelines.
  Arms: Experimental group
Procedure: RARP+ePLND — Participants will undergo robot-assisted radical prostatectomy (RARP) with extended pelvic lymph node dissection (ePLND), encompassing bilateral removal of obturator, external iliac, internal iliac, and common iliac lymph nodes. The dissection field extends laterally to the genitofemoral nerve, medially to the bladder wall, proximally to the ureter crossing the common iliac vessels, and distally to the deep circumflex iliac vein and femoral canal.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to evaluate efficacy and safety of radical prostatectomy (RP) with or without salvage radiotherapy versus RP with extended pelvic lymph node dissection (ePLND) in males who have localized intermediate/high-risk prostate cancer with a Briganti nomogram no less than 7%. The main questions this study aim to answer are:

1. Is RP with or without salvage radiotherapy non-inferior to RP with ePLND in efficacy for patients with localized intermediate/high-risk prostate cancer with a Briganti nomogram no less than 7%?
2. Will complication rates of RP with or without salvage radiotherapy be significantly lower than those of RP with ePLND?

Researchers will compare the experimental arm (robot-assisted laparoscopic radical prostatectomy with or without salvage radiotherapy) versus the control arm (robot-assisted laparoscopic radical prostatectomy with ePLND) to see if differences exist in oncological efficacy and safety outcomes.

Participants will:

1. Undergo one of the following surgical interventions:

   1. Robot-assisted laparoscopic radical prostatectomy (RARP) with extended pelvic lymph node dissection (ePLND), OR
   2. RARP alone, followed by salvage radiotherapy only if biochemical recurrence occurs postoperatively
2. Complete scheduled monitoring activities:

   1. Serum PSA testing: Monthly or every 3 months within 2 years after surgery
   2. PSMA PET/CT scans: Annually until study completion
   3. Report all treatment-related complications within 24 hours of onset

ELIGIBILITY:
Inclusion Criteria:

* Provided signed and dated informed consent form.
* Be male aged 18-80 years at consent.
* Commit to protocol compliance and complete all study procedures.
* Medically fit to tolerate interventions, including PSMA PET imaging, RARP, pelvic radiotherapy.
* Diagnosis of localized intermediate/high-risk prostate cancer (miN0M0):

  i. Confirmed by: systematic biopsy + PSA + PSMA PET/MRI. ii. Briganti nomogram (2017)≥7%. iii. Candidate for radical prostatectomy. iv. D'Amico:
  1. Intermediate-risk: PSA 10-20ng/mL OR Gleason 7 (ISUP Grade 2/3) OR cT2b;
  2. High-risk: PSA>20ng/mL OR Gleason>7 (ISUP Grade 4/5) OR cT2c.

     Exclusion Criteria:
* Prior treatments for prostate cancer, including radiotherapy, chemotherapy or endocrine therapy.
* Non-acinar adenocarcinoma histology on biopsy.
* Preoperative evidence of metastasis: nodal(N1), locally advanced(T3-4), or distant(M1) disease on imaging.
* History of pelvic lymphadenectomy or radiotherapy.
* Other malignancies within 5 years.
* Contraindications to radical prostatectomy or being deemed surgically inoperable upon clinical assessment.
* Contraindications to radiotherapy or intolerance determined by radiation oncologists.
* Severe allergy to PSMA PET ligands or excipients.
* Any other conditions precluding PSMA PET examination.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
2-year Biochemical-recurrence Free Survival rate (2-year BFS) | 2 years from randomization
  The 2-year biochemical recurrence-free survival rate (2-year BFS) will be recorded from randomization. Biochemical recurrence (BCR) is defined as serum PSA≥0.2ng/mL confirmed by at least one repeat test >6 weeks postoperatively. Time to first BCR event is measured:
  1. For control group: After RARP completion.
  2. For experimental group: After salvage radiotherapy completion.

SECONDARY OUTCOMES:
PSA doubling time, PSADT | baseline and 2 years
Radiographic progression-free survival, rPFS | 2 years from randomization
Time to First biochemical recurrence (BCR) event in the experimental group | 2 years from randomization
Overall survival, OS | 2 years from randomization

OTHER OUTCOMES:
Operative time | Perioperative
Incidence Rate and Severity of Radiation-related complications | From radiotherapy initiation through 1 month post-treatment
  1. Radiation proctitis
  2. Radiation cystitis Complications will be categorized per CTCAE v5.0, with Grade ≥3 defined as clinically significant.
Incidence Rate and Severity of Intraoperative and 30-day postoperative complications | During index hospitalization (up to 30 days post-op)
  1. lymphatic leakage
  2. lymphocele
  3. prolonged pelvic drainage (>2 weeks)
  4. obturator nerve injury
  5. pelvic organ injury (rectum/bladder/vasculature/ureter)
  6. acute urinary retention
  Complications will be categorized per CTCAE v5.0, with Grade ≥3 defined as clinically significant.
Intraoperative blood loss | Perioperative
Hospital stay length | Perioperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No